CLINICAL TRIAL: NCT01981044
Title: A SERI® Surgical Scaffold Postmarket Study of Soft Tissue Support in Ventral Hernia Repair
Brief Title: SERI® Surgical Scaffold Postmarket Study of Soft Tissue Support in Ventral Hernia Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty accruing patients; business decision
Sponsor: Sofregen Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURE-007
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Results first posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Ventral Hernia Repair

ARMS (1):
- SERI® Surgical Scaffold (Experimental): It is a prospective, multicenter, single-arm, post-market on-label clinical study of a 510(k)-cleared device.
  Interventions: Device: Silk surgical mesh

INTERVENTIONS:
Device: Silk surgical mesh — A CE Marked, 510(k) cleared, knitted, multi-filament, bioengineered, silk mesh indicated for use as a transitory scaffold for soft tissue support and repair
  Other Names: SERI® Surgical Scaffold

SUMMARY:
Prospective, multi center, single arm, clinical study to obtain clinical experience with the use of SERI® Surgical Scaffold for soft tissue support in ventral hernia repair.

DETAILED DESCRIPTION:
Prospective, multicenter, single-arm, post-market on-label clinical study of a 510(k)-cleared device. Subjects will be followed for 24 months post SERI placement during index hernia repair surgery. Study visits will occur at screening, from SERI implantation through hospital discharge and then post SERI implantation at month(s) 1, 3, 6, 12, 18, and 24 for all enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

The following are requirements for entry into the study. The subject MUST:

1. Be ≥ 18 years of age

2. Be diagnosed with a ventral hernia as defined as:

1. Midline Ventral Hernia AND
2. Defect(s) MUST meet the following criteria:

   * contained within an anatomical area of ≤ 150 cm2
   * not be longer than 8cm in any direction
   * size must have a total sum ≤ 64 cm2
3. Be eligible for retro-rectus placement of SERI
4. Have a BMI < 40

Exclusion Criteria:

The following are criteria for exclusion from participating in the study. The subject must

NOT:

1. Be > 70 years of age
2. Have prior occurrence of ventral hernia or parastomal hernia
3. Have a presence of a stoma or have a perforated bowel
4. Have any documented disease which is clinically known to impact wound healing, including Chronic Obstructive Pulmonary Disease (COPD), and Congestive Heart Failure (CHF), with the exception of controlled diabetes
5. Have documented history of diabetes with an A1C of ≥ 8 at time of pre-operative visit
6. Have documented autoimmune disease, an immune deficiency, or be on immunosuppressive drugs with the exception of steroids for:

1. prophylactic one-time-use administered peri-operatively

2. inhaled general use

3. topical administration

7. Have documented collagen-vascular, connective tissue, bleeding disorders and/or on anticoagulation therapy, with the exception of baby aspirin for one week prior to SERI placement

8. Have documented cancer < 6 months prior to surgery or chemotherapy treatment < 6 months prior to surgery

9. Have documented history of abdominal radiation therapy or is expected to have abdominal radiation therapy during the conduct of this study

10. Have documented history of liver disease and/or renal failure requiring dialysis

11. Have documented history of a previous wound infection at the surgical site or have an active infection at the time of surgery

12. Have had prior surgery with synthetic and/or biologic mesh in the abdominal, chest or pelvic area

13. Have documented allergy to silk

14. Have documented UTI at the time of surgery

15. Have smoked within 6 weeks of surgery and have a positive nicotine test at time of preoperative visit

16. Have a concurrent procedure intra-operatively (with the exception of lysis of abdominal adhesions)

17. Require intra-peritoneal or bridging placement of the soft tissue support device or require component separation at time of surgery

18. Have surgical circumstances that are contraindicated for use of SERI™ Surgical Scaffold per the supplied package insert

19. Have a concomitant unrelated condition of abdominal/chest wall/skin that would require a surgical intervention during the follow-up period

20. Have documented alcohol and/or substance abuse problem at time of pre-operative visit

21. Be pregnant, lactating, or if of childbearing potential, be unwilling to use contraceptive methods and avoid pregnancy throughout the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2015-09-25 (Actual); Study Completion 2016-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan Medical
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SERI® Surgical Scaffold
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SERI® Surgical Scaffold
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Hernia Recurrence
Description: Hernia recurrence at 6 months post-operatively will be assessed by the Investigator and then confirmed via an independent physician.
Time Frame: 6 months postoperatively
Population: Adults between 18 and 70 years of age with SERI for ventral hernia repair
Measure: Count of Participants; unit: Participants
Arm/Group | SERI® Surgical Scaffold
Number analyzed (Participants) | 1
Participants
  Intact primary hernia repair with SERI | 1
  Hernia reoccurred | 0

2. Primary Outcome: Rate of Hernia Recurrence
Description: Hernia recurrence at 12 months post-operatively will be assessed by the Investigator and then confirmed via an independent physician.
Time Frame: 12 months postoperatively
Population: Adults between 18 and 70 years of age using SERI for ventral hernia repair
Measure: Count of Participants; unit: Participants
Arm/Group | SERI® Surgical Scaffold
Number analyzed (Participants) | 1
Participants
  Intact primary hernia repair | 1
  Hernia reoccurred | 0

3. Primary Outcome: Rate of Hernia Recurrence
Description: Hernia recurrence at 24 months post-operatively will be assessed by the Investigator and then confirmed via an independent physician.
Time Frame: 24 months postoperatively
Population: Adults between 18 and 70 years of age with SERI for ventral hernia repair
Measure: Count of Participants; unit: Participants
Arm/Group | SERI® Surgical Scaffold
Number analyzed (Participants) | 1
Participants
  Intact primary repair with SERI | 1
  Hernia reoccurrence | 0

ADVERSE EVENTS:
Time Frame: 24 months after the ventral hernia repair procedure
Description: AE definitions consistent with clinicaltrials.gov
  Throughout the course of the study, AEs will be monitored and reported in an AE eCRF, including seriousness, severity, relationship to device, and action taken. If AEs occur, the first concern will be the safety of the study participants. The Investigator and the research staff will monitor each subject closely, and, should a complication occur, they will use their medical judgment to do whatever is necessary to treat the problem.
Arm/Group | SERI® Surgical Scaffold
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SERI® Surgical Scaffold (N=1)
Abcess (Skin and subcutaneous tissue disorders) | 1 (4)
Fluid Collection (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SERI® Surgical Scaffold (N=1)
Pain (Skin and subcutaneous tissue disorders) | 1 (3)
Abdominal Muscle Spasm (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No